CLINICAL TRIAL: NCT02273947
Title: An Open-Label, Randomized, Crossover Adaptive Design Study to Assess the Effect of Food on the Pharmacokinetics of BMS-955176 Administered as a Micronized Crystalline Tablet in Healthy Subjects
Brief Title: Food Effect Study With BMS-955176
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 206221
Record Dates: First submitted 2014-10-10; First posted 2014-10-24 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — BMS-955176

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (21):
- Arm 1 (ABDC): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment as specified
  Interventions: Drug: BMS-955176
- Arm 2 (BCAD): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment as specified
  Interventions: Drug: BMS-955176
- Arm 3 (CDBA): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment as specified
  Interventions: Drug: BMS-955176
- Arm 4 (DACB): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment as specified
  Interventions: Drug: BMS-955176
- Arm 5 (EFHG): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment as specified
  Interventions: Drug: BMS-955176
- Arm 6 (FGEH): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment as specified
  Interventions: Drug: BMS-955176
- Arm 7 (GHFE): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment as specified
  Interventions: Drug: BMS-955176
- Arm 8 (HEGF): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment as specified
  Interventions: Drug: BMS-955176
- Arm 9 (IJK): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176
- Arm 10 (JKI): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176
- Arm 11 (KIJ): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176
- Arm 12 (IKJ): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176
- Arm 13 (JIK): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176
- Arm 14 (KJI): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176
- Arm 15 (LMN): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176
- Arm 16 (OPQ): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176
- Arm 17 (PQO): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176
- Arm 18 (QOP): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176
- Arm 19 (OQP): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176
- Arm 20 (POQ): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176
- Arm 21 (QPO): BMS-955176 (Experimental): BMS-955176 single dose by mouth for each treatment specified
  Interventions: Drug: BMS-955176

INTERVENTIONS:
Drug: BMS-955176 — Single dose by mouth for each treatment specified

SUMMARY:
The purpose of this study is to assess the impact of a light meal, a standard meal, and a high fat meal on the PK of BMS-955176 MC tablet at a dose of 180 mg, relative to fasted conditions.

DETAILED DESCRIPTION:
Primary Purpose

Other: This study will assess the impact of a light meal, a standard meal, and a high fat meal on the pharmacokinetics (PK) of BMS-955176 micronized crystalline (MC) tablet at a dose of 180 mg relative to fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examinations, vital sign measurements, 12-lead ECG measurements, and clinical laboratory test results
* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive. BMI = Weight (kg)/[Height (m)]2
* Men and women, ages 18 to 50 years, inclusive
* Women must not be of childbearing potential, must not be breastfeeding

Exclusion Criteria:

* Any significant acute or chronic medical illness
* History of cardiac disease or clinically significant cardiac arrhythmias
* Current or recent (within 3 months of study drug administration) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* Any gastrointestinal surgery (including cholecystectomy) that could impact upon the absorption of study drug

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) for BMS-955176 | Up to Day 4 of Period 4
Area under the plasma concentration-time curve from time zero to 72 hours post-dose [AUC(0-72)] for BMS-955176 | Up to Day 4 of Period 4
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] for BMS-955176 | Up to Day 4 of Period 4
Plasma concentration at 24 hours post-dose (C24) for BMS-955176 | Up to Day 4 of Period 4

SECONDARY OUTCOMES:
Safety and tolerability | Up to 30 days post discontinuation of dosing
  Safety and tolerability measured by incidence of AEs, serious AEs (SAEs), AEs leading to discontinuation and death, marked abnormalities in clinical laboratory tests, viral sign measurements, ECGs, and physical examination Adverse Events (AEs), Electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Ruddington Fields, Nottinghamshire, United Kingdom